CLINICAL TRIAL: NCT05763446
Title: Predictive Factors for Massive Transfusion During Liver Transplantation: an Observational Study
Brief Title: Predictive Factors for Massive Transfusion During Liver Transplantation
Acronym: TRADIFEG
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4216
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Liver Transplant; Complications
Keywords: Transfusions; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplantation (LT) is the treatment of choice for patients with end-stage liver disease (1). LT is often associated with severe intraoperative blood loss and the literature has had a great interest in clarifying the predictive factors for transfusion requirements during this surgery. Despite the advances in surgical techniques, graft preservation, and anesthetic management achieved over the past two decades, intraoperative bleeding and blood component consumption during LT are still issues of current interest. The requirement for blood components is highly variable between different transplant centers and ranges from none to many units of red blood cells (RBC), plasma, and platelets per patient. Bleeding associated with LT is multifactorial. Among the pre-transplantation factors, portal hypertension and coagulation defects are of great importance. The latter can develop or amplify during the anaepatic and/or neohepatic phase due to the absence of hepatic metabolic function, hyperfibrinolysis or platelet sequestration in the graft. In the literature, the higher transfusion requirement (HTR) is associated with worse postoperative outcomes, with an increase in both the length of stay in the intensive care unit (ICU) and in hospital, and mortality.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the influence of increased transfusion requirements on the prognosis of patients undergoing LT and the risk factors for HTR. HTR is defined as the consumption of packed red blood cells (GRC) ≥ 5 units in the first 24 hours of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation

Exclusion Criteria:

* Age <18 years
* Retransplantation within 30 days
* Combined kidney-liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  90-day postoperative mortality after liver transplantation

SECONDARY OUTCOMES:
Postoperative mechanical ventilation | 48 hours
  Duration of invasive mechanical ventilation
Intensive care unit stay | Days until discharge from ICU, an average of 5 days
  Duration of intensive care unit stay
In-hospital stay | Days until discharge from the hospital, an average of 14 days
  Hospital stay duration after liver transplant
Post-transplant complication | 90 days
  90-day postoperative complications after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Paola Aceto, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - UOC Anestesia delle Chirurgie Generali e dei Trapianti, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome